CLINICAL TRIAL: NCT05831072
Title: Efficacy of Mindfulness-cognitive Oriented Group Intervention Program on Depressive Symptoms, Coping Strategies and Quality of Life in University Students
Brief Title: Efficacy of Mindfulness-cognitive Oriented Group Intervention Program on Depressed University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Yun-Ling Chen, Assistant Professor, Chung Shan Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS1-22140
Record Dates: First submitted 2023-03-02; First posted 2023-04-26 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Depression in Adolescence
Keywords: mindfulness-based cognitive therapy; depressive symptoms; coping strategy; quality of life; university students
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Students who have suitable cognitive capacity and minor and above level of depressive symptoms will be included in the study. Each single group will be 16 students or below.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness-cognitive oriented group (Experimental): Participants will receive a 4-week intervention of mindfulness-cognitive oriented group program.
  Interventions: Behavioral: Mindfulness-cognitive oriented group program

INTERVENTIONS:
Behavioral: Mindfulness-cognitive oriented group program — Mindfulness-cognitive oriented group program is a 4-week program based on the theory of mindfulness-based cognitive therapy (MBCT). The main elements of MBCT such as mindfulness breathing, raisin meditation for mindful eating, body scan and mindfulness walking are included. In addition to the weekly intervention, participants are also required to do the mindfulness practice at home.

SUMMARY:
The goal of this study is to reduce depressive symptoms as well as increase the positive coping strategy and quality of life in depressed university students. The main question it aims to answer is:

• The efficacy of 4-week mindfulness-cognitive oriented group program

The participants will be requested to participate in a 4-week program and do the mindfulness practice at home.

DETAILED DESCRIPTION:
In this study, the investigators will recruit university students through a poster at Chung Shan Medical University and the Internet.

For the screening, students will be requested to complete the assessments of the Saint Louis University Mental Status and Beck Depression Inventory-II. Students who have suitable cognitive capacity and minor and above level of depressive symptoms will be included in the study. The participants will receive a mindfulness-cognitive oriented group program for 4 weeks.

All the subjects will fill out the self-reported questionnaires at baseline, after the intervention, and one-month after the intervention. The assessments include Beck Depression Inventory-II, Brief Coping Orientation to Problems Experienced Inventory, World Health Organization Quality-of-Life Scale-BREF, Occupational Balance Questionnaire, Role Checklist, and Occupational Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* currently enrolled as a student at Chung Shan Medical University
* between 18 and 30 years old
* The Saint Louis University Mental Status (SLUMS) total score is greater than 26
* the total score of Beck Depression Inventory-II (BDI-II) Chinese version is above 13
* fluency in spoken Mandarin

Exclusion Criteria:

* the score of item 9 (suicidal ideation) of Beck Depression Inventory-II (BDI-II) Chinese version > 0
* a current diagnosis of depressive disorder
* a current diagnosis of a major physical illness (e.g., cancer, cerebrovascular disease (stroke), spinal cord injury, congenital or genetic disease, chronic renal failure, autoimmune disease, burns) or psychological disease (psychotic or other psychiatric disorders, bipolar disorder, substance-related or addiction disorder, neurodevelopmental disorder, neurocognitive disorder, substance- or drug-induced depression)
* currently taking psychiatric medication or receiving psychotherapy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
Depression (screening) | screening
  Beck Depression Inventory - II (BDI-II) contains 21 items (each of them is scored on a scale of 0-3) in order to measure the depressive symptoms of participants. Higher scores indicates greater level of depression. 0-13 is considered a none or minimal, 14-19 is mild, 20-28 is moderate, and 29-63 is severe level of depression.
Depression (baseline) | baseline
  Beck Depression Inventory - II (BDI-II) contains 21 items (each of them is scored on a scale of 0-3) in order to measure the depressive symptoms of participants. Higher scores indicates greater level of depression. 0-13 is considered a none or minimal, 14-19 is mild, 20-28 is moderate, and 29-63 is severe level of depression.
Depression (post-intervention) | post-intervention (up to 4 weeks)
  Beck Depression Inventory - II (BDI-II) contains 21 items (each of them is scored on a scale of 0-3) in order to measure the depressive symptoms of participants. Higher scores indicates greater level of depression. 0-13 is considered a none or minimal, 14-19 is mild, 20-28 is moderate, and 29-63 is severe level of depression.
Depression (follow-up) | 1-month follow-up
  Beck Depression Inventory - II (BDI-II) contains 21 items (each of them is scored on a scale of 0-3) in order to measure the depressive symptoms of participants. Higher scores indicates greater level of depression. 0-13 is considered a none or minimal, 14-19 is mild, 20-28 is moderate, and 29-63 is severe level of depression.
Coping style (baseline) | baseline
  Brief Coping Orientation to Problems Experienced Inventory (Brief COPE) is a 28-item self-report questionnaire that using a 4-point rating scale in each item. It determines individual's primary coping styles with stressful life event, including approaching coping strategy, positive avoiding coping strategy and negative avoiding coping strategy. Scores are presented for three overarching coping styles as average scores, indicating the degree to which the respondent has been engaging in that coping style.
Coping style (post-intervention) | post-intervention (up to 4 weeks)
  Brief Coping Orientation to Problems Experienced Inventory (Brief COPE) is a 28-item self-report questionnaire that using a 4-point rating scale in each item. It determines individual's primary coping styles with stressful life event, including approaching coping strategy, positive avoiding coping strategy and negative avoiding coping strategy. Scores are presented for three overarching coping styles as average scores, indicating the degree to which the respondent has been engaging in that coping style.
Coping style (follow-up) | 1-month follow-up
  Brief Coping Orientation to Problems Experienced Inventory (Brief COPE) is a 28-item self-report questionnaire that using a 4-point rating scale in each item. It determines individual's primary coping styles with stressful life event, including approaching coping strategy, positive avoiding coping strategy and negative avoiding coping strategy. Scores are presented for three overarching coping styles as average scores, indicating the degree to which the respondent has been engaging in that coping style.
Quality of life (baseline) | baseline
  The World Health Organization Quality-of-Life Scale (WHOQOL-BREF) is a 28-item self-report questionnaire with a five point rating scale for each item (from 1 to 5). There are four domains in WHOQOL-BREF, including physical health, psychological health, social relationships, and environment. A higher score indicates a higher quality of life.
Quality of life (post-intervention) | post-intervention (up to 4 weeks)
  The World Health Organization Quality-of-Life Scale (WHOQOL-BREF) is a 28-item self-report questionnaire with a five point rating scale for each item (from 1 to 5). There are four domains in WHOQOL-BREF, including physical health, psychological health, social relationships, and environment. A higher score indicates a higher quality of life.
Quality of life (follow-up) | 1-month follow-up
  The World Health Organization Quality-of-Life Scale (WHOQOL-BREF) is a 28-item self-report questionnaire with a five point rating scale for each item (from 1 to 5). There are four domains in WHOQOL-BREF, including physical health, psychological health, social relationships, and environment. A higher score indicates a higher quality of life.

SECONDARY OUTCOMES:
Occupational balance (baseline) | baseline
  Occupational Balance Questionnaire (OBQ) is a 11-item questionnaire with a four point response scale for each item (from 0 to 3) by the level of agreemtent with each of the affirmations. The OBQ is used to measure the perception of current occupational balance in daily life. The total score is ranged from 0 to 33. A higher score indicates a greater occupational balance.
Occupational balance (post-intervention) | post-intervention (up to 4 weeks)
  Occupational Balance Questionnaire (OBQ) is a 11-item questionnaire with a four point response scale for each item (from 0 to 3) by the level of agreemtent with each of the affirmations. The OBQ is used to measure the perception of current occupational balance in daily life. The total score is ranged from 0 to 33. A higher score indicates a greater occupational balance.
Occupational balance (follow-up) | 1-month follow-up
  Occupational Balance Questionnaire (OBQ) is a 11-item questionnaire with a four point response scale for each item (from 0 to 3) by the level of agreemtent with each of the affirmations. The OBQ is used to measure the perception of current occupational balance in daily life. The total score is ranged from 0 to 33. A higher score indicates a greater occupational balance.
Role checklist (baseline) | baseline
  Role checklist is used to assess the major roles that organize participant's daily life and the value of each role. The roles included the student, worker, volunteer, caregiver, home maintainer, friend, family member, religious participant, hobbyist, and participant in organizations. A higher number of roles means participating more roles in daily life. A higher score in the value of roles means more productive behaviors participants needed or desired.
Role checklist (post-intervention) | post-intervention (up to 4 weeks)
  Role checklist is used to assess the major roles that organize participant's daily life and the value of each role. The roles included the student, worker, volunteer, caregiver, home maintainer, friend, family member, religious participant, hobbyist, and participant in organizations. A higher number of roles means participating more roles in daily life. A higher score in the value of roles means more productive behaviors participants needed or desired.
Role checklist (follow-up) | 1-month follow-up
  Role checklist is used to assess the major roles that organize participant's daily life and the value of each role. The roles included the student, worker, volunteer, caregiver, home maintainer, friend, family member, religious participant, hobbyist, and participant in organizations. A higher number of roles means participating more roles in daily life. A higher score in the value of roles means more productive behaviors participants needed or desired.
Occupational questionnaire (baseline) | baseline
  Occupational questionnaire (OQ) is used to record daily occupations on 30-minute interval for a typical day. Each activity need to be classified as work, activity of daily living, recreation or rest and be rated for the competence, value, and interest using a five point rating scale. It indicates how well the participants do the activity, how important the activity is as well as how enjoyable the activity is. The higher score means better satisfaction, value and enjoyment of activity that the participant did.
Occupational questionnaire (post-intervention) | post-intervention (up to 4 weeks)
  Occupational questionnaire (OQ) is used to record daily occupations on 30-minute interval for a typical day. Each activity need to be classified as work, activity of daily living, recreation or rest and be rated for the competence, value, and interest using a five point rating scale. It indicates how well the participants do the activity, how important the activity is as well as how enjoyable the activity is. The higher score means better satisfaction, value and enjoyment of activity that the participant did.
Occupational questionnaire (follow-up) | 1-month follow-up
  Occupational questionnaire (OQ) is used to record daily occupations on 30-minute interval for a typical day. Each activity need to be classified as work, activity of daily living, recreation or rest and be rated for the competence, value, and interest using a five point rating scale. It indicates how well the participants do the activity, how important the activity is as well as how enjoyable the activity is. The higher score means better satisfaction, value and enjoyment of activity that the participant did.

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Ling Chen, Doctor, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cladder-Micus MB, Speckens AEM, Vrijsen JN, T Donders AR, Becker ES, Spijker J. Mindfulness-based cognitive therapy for patients with chronic, treatment-resistant depression: A pragmatic randomized controlled trial. Depress Anxiety. 2018 Oct;35(10):914-924. doi: 10.1002/da.22788. Epub 2018 Aug 8. PMID 30088834
- [Result] Compas BE, Connor-Smith JK, Saltzman H, Thomsen AH, Wadsworth ME. Coping with stress during childhood and adolescence: problems, progress, and potential in theory and research. Psychol Bull. 2001 Jan;127(1):87-127. PMID 11271757
- [Result] Demarzo M, Montero-Marin J, Puebla-Guedea M, Navarro-Gil M, Herrera-Mercadal P, Moreno-Gonzalez S, Calvo-Carrion S, Bafaluy-Franch L, Garcia-Campayo J. Efficacy of 8- and 4-Session Mindfulness-Based Interventions in a Non-clinical Population: A Controlled Study. Front Psychol. 2017 Aug 8;8:1343. doi: 10.3389/fpsyg.2017.01343. eCollection 2017. PMID 28848465
- [Result] Farb N, Anderson A, Ravindran A, Hawley L, Irving J, Mancuso E, Gulamani T, Williams G, Ferguson A, Segal ZV. Prevention of relapse/recurrence in major depressive disorder with either mindfulness-based cognitive therapy or cognitive therapy. J Consult Clin Psychol. 2018 Feb;86(2):200-204. doi: 10.1037/ccp0000266. Epub 2017 Dec 21. PMID 29265831
- [Result] Foroughi A, Sadeghi K, Parvizifard A, Parsa Moghadam A, Davarinejad O, Farnia V, Azar G. The effectiveness of mindfulness-based cognitive therapy for reducing rumination and improving mindfulness and self-compassion in patients with treatment-resistant depression. Trends Psychiatry Psychother. 2020 Jun;42(2):138-146. doi: 10.1590/2237-6089-2019-0016. Epub 2020 Jul 17. PMID 32696895
- [Result] Kuyken W, Byford S, Taylor RS, Watkins E, Holden E, White K, Barrett B, Byng R, Evans A, Mullan E, Teasdale JD. Mindfulness-based cognitive therapy to prevent relapse in recurrent depression. J Consult Clin Psychol. 2008 Dec;76(6):966-78. doi: 10.1037/a0013786. PMID 19045965
- [Result] Musa ZA, Soh KL, Mukhtar F, Soh KY, Oladele TO, Soh KG. Impact of Mindfulness-Based Cognitive Therapy on Depressive Symptoms Reduction among Depressed Patients in Nigeria: A Randomized Controlled Trial. Issues Ment Health Nurs. 2021 Jul;42(7):667-675. doi: 10.1080/01612840.2020.1821139. Epub 2020 Sep 30. PMID 32996802
- [Result] Probst T, Schramm E, Heidenreich T, Klein JP, Michalak J. Patients' interpersonal problems as moderators of depression outcomes in a randomized controlled trial comparing mindfulness-based cognitive therapy and a group version of the cognitive-behavioral analysis system of psychotherapy in chronic depression. J Clin Psychol. 2020 Jul;76(7):1241-1254. doi: 10.1002/jclp.22931. Epub 2020 Jan 30. PMID 31997369
- [Result] Ritvo P, Knyahnytska Y, Pirbaglou M, Wang W, Tomlinson G, Zhao H, Linklater R, Bai S, Kirk M, Katz J, Harber L, Daskalakis Z. Online Mindfulness-Based Cognitive Behavioral Therapy Intervention for Youth With Major Depressive Disorders: Randomized Controlled Trial. J Med Internet Res. 2021 Mar 10;23(3):e24380. doi: 10.2196/24380. PMID 33688840
- [Result] Schanche E, Vollestad J, Visted E, Svendsen JL, Osnes B, Binder PE, Franer P, Sorensen L. The effects of mindfulness-based cognitive therapy on risk and protective factors of depressive relapse - a randomized wait-list controlled trial. BMC Psychol. 2020 Jun 5;8(1):57. doi: 10.1186/s40359-020-00417-1. PMID 32503649
- [Result] Segal ZV, Dimidjian S, Beck A, Boggs JM, Vanderkruik R, Metcalf CA, Gallop R, Felder JN, Levy J. Outcomes of Online Mindfulness-Based Cognitive Therapy for Patients With Residual Depressive Symptoms: A Randomized Clinical Trial. JAMA Psychiatry. 2020 Jun 1;77(6):563-573. doi: 10.1001/jamapsychiatry.2019.4693. PMID 31995132
- [Result] Sun Y, Li Y, Wang J, Chen Q, Bazzano AN, Cao F. Effectiveness of Smartphone-Based Mindfulness Training on Maternal Perinatal Depression: Randomized Controlled Trial. J Med Internet Res. 2021 Jan 27;23(1):e23410. doi: 10.2196/23410. PMID 33502326
- [Result] Winnebeck E, Fissler M, Gartner M, Chadwick P, Barnhofer T. Brief training in mindfulness meditation reduces symptoms in patients with a chronic or recurrent lifetime history of depression: A randomized controlled study. Behav Res Ther. 2017 Dec;99:124-130. doi: 10.1016/j.brat.2017.10.005. Epub 2017 Oct 12. PMID 29078199
- [Result] Zemestani M, Fazeli Nikoo Z. Effectiveness of mindfulness-based cognitive therapy for comorbid depression and anxiety in pregnancy: a randomized controlled trial. Arch Womens Ment Health. 2020 Apr;23(2):207-214. doi: 10.1007/s00737-019-00962-8. Epub 2019 Apr 13. PMID 30982086